CLINICAL TRIAL: NCT00003001
Title: Phase I/II Study of 5-Fluorouracil/Folinic Acid/Gemcitabine in Patients With Advanced Colorectal Carcinoma
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent or Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Stony Brook University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065561; SUNY-HSC-97-2824; NCI-V97-1256
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2002-04

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Gemcitabine; Leucovorin

INTERVENTIONS:
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combination chemotherapy consisting of fluorouracil, leucovorin, and gemcitabine in treating patients with recurrent or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate and survival of patients with recurrent or metastatic colorectal carcinoma treated with fluorouracil (5-FU), leucovorin calcium, and gemcitabine. II. Evaluate and establish the toxic effect profile of 5-FU, leucovorin calcium, and gemcitabine in these patients.

OUTLINE: This is a dose escalation study. Patients receive intravenous leucovorin calcium for 60 minutes and bolus infusions of fluorouracil (5-FU), followed by gemcitabine infusions, weekly for six weeks followed by 2 weeks of rest. The dosage of gemcitabine is increased if fewer than 3 of the first 6 patients experience grade 3-4 toxicities. Phase II proceeds at the maximum tolerated dose (1 dose level below that at which 3 patients experience grade 3-4 toxicities). Patients receive a minimum of two courses of treatment to be considered evaluable for response. Patients with stable disease, partial, or complete remission may continue therapy for up to six treatment cycles. Patients exhibiting disease progression or intolerable toxic effects are removed from the study.

PROJECTED ACCRUAL: A total of 63 patients will be accrued.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or metastatic primary colorectal carcinoma Must have measurable disease (evaluable disease acceptable in Phase I)

PATIENT CHARACTERISTICS: Age: Not specified Performance Status: ECOG 0-3 Life Expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL OR 3.0 mg/dL in patients with liver metastases Liver enzymes no greater than 3.0 times upper limit of normal (in patients with liver metastases) Renal: Not specified Other: Not pregnant or lactating Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Prior chemotherapy for metastatic disease allowed Prior treatment with 5-FU allowed Prior treatment with irinotecan allowed Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy (measurable disease must be located outside the prior radiotherapy portal) Surgery: Not specified Other: Prior treatment with folinic acid allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 1997-04

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Madajewicz, MD, PhD, Study Chair — Stony Brook University
Locations (1):
- State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York, United States